CLINICAL TRIAL: NCT01399645
Title: Randomized Trial of Liraglutide and Insulin Therapy on Hepatic Steatosis as Measured by MRI and MRS in Metformin-treated Patients With Type 2 Diabetes: an Open Pilot Study
Brief Title: Study of Liraglutide Versus Insulin on Liver Fat Fraction in Patients With Type 2 Diabetes
Acronym: LIRAINS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); Diabetes Québec (Other); Radiological Society of North America (Other); Canadian Heads of Academic Radiology-GE Healthcare Development Award (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE09.159
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis; Type 2 Diabetes
Keywords: Randomized trial; Open label; Pilot study; Single center
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Insulin Glargine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide-Metformin (Experimental): Liraglutide (Victoza, Novo Nordisk) at a dose of 0.6 - 1.8 mg subcutaneous per day until the end of the study.
  All subjects will be given metformin with a starting dose of 500 mg in one tablet twice daily given before or during meals for the duration of the study.
  Interventions: Drug: Liraglutide-metformin vs insulin-metformin
- Insulin-Metformin (Experimental): Insulin glargine (Lantus, Sanofi-Aventis) with an initial bedtime starting dose of 10 IU. The patients will be taught to increase their insulin dose by 1 unit each day until achieving an FPG ≤ 7.0 mmol/L.
  All subjects will be given metformin with a starting dose of 500 mg in one tablet twice daily given before or during meals for the duration of the study.
  Interventions: Drug: Liraglutide-metformin vs insulin-metformin

INTERVENTIONS:
Drug: Liraglutide-metformin vs insulin-metformin — Liraglutide (Victoza, Novo Nordisk) at a dose of 0.6 - 1.8 mg subcutaneous per day.
  Insulin glargine (Lantus, Sanofi-Aventis) with an initial bedtime starting dose of 10 IU.
  Other Names: Liraglutide; Victoza; Insulin glargine; Lantus

SUMMARY:
This study is conducted to test the hypothesis that in type 2 diabetic adults with fatty liver who are resistant to metformin, treatment with liraglutide in combination with metformin will cause an absolute reduction in liver fat superior to insulin-metformin treatment within a 3-month period, as measured by magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Background: Non-alcoholic fatty liver disease (NAFLD) can now be identified in 70% of patients with type 2 diabetes. Insulin can be introduced at any point in the treatment of diabetes, but is potentially lipogenic. Preliminary studies have shown conflicting results on the impact of insulin on fatty liver.

Objectives: This study is conducted to test the hypothesis that in type 2 diabetic adults with NAFLD who are resistant to metformin, treatment with liraglutide in combination with metformin will cause an absolute reduction in liver fat superior to insulin-metformin treatment within a 3-month period, as measured by in vivo MRI and MRS.

Design: This will be a prospective, open label, randomized parallel trial to evaluate whether 12 weeks of treatment with a) liraglutide-metformin will improve steatosis in type 2 diabetic adults with NAFLD compared to treatment with b) insulin-metformin. Before and post-treatment MRI and MRS will be read blindly for quantification of steatosis. The primary outcome measure is defined as an improvement in steatosis of 5% before and after treatment between the 2 treatment groups.

Methods: Thirty-six patients will be randomized to either study group. After baseline metabolic measurements by blood sampling, transient ultrasound elastography, MRI and MRS, all subjects will be given metformin with a starting dose of 500 mg in one tablet twice daily. In addition, patients will be randomized to receive either liraglutide (0.6 - 1.8 mg subcutaneous per day ) or insulin glargine with an initial bedtime starting dose of 10 IU for a duration of 3 months.

Expected results: The results of this study will provide preliminary data for a large scale study comparing the 2 therapeutic regimen and establish the utility of MRI and MRS to monitor medical treatment in diabetic patients with fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 y.o. or older at screening (first visit),
* Are ambulatory,
* Are known for type 2 diabetes with criteria of failure of metformin monotherapy, metformin-sulfonylurea, metformin-repaglinide combined therapy defined as HbA1C ≥6.5,
* Abdominal girth > 94 cm for men and > 80 cm for women,
* Understand French or English instruction,
* Able to comprehend and willingness to provide voluntary consent.

Exclusion Criteria:

* Have any contra-indications for MRI (such as metallic implants, pacemaker or claustrophobia),
* Have type 1 diabetes or have had episodes of ketoacidosis,
* Have any major debilitating disease including malignant disorders,
* Have had, within the last 6 months, evidence of significant heart disease or stroke, including myocardial infarction, unstable angina, coronary bypass and/or percutaneous transluminal coronary angioplasty (PTCA), congestive heart failure (New York Heart Association Class III-IV), or severe ischemic disease,
* Patients having received insulin within 3 months prior to screening,
* Have a serum creatine above >150 mmol/L or estimated GFR < 30 mL/min,
* Women seeking pregnancy,
* Have a history of chronic liver disease other than NAFLD, including HBV and HCV infection, hemochromatosis, Wilson's disease, alpha-1-antitrypsin deficiency, autoimmune hepatitis,
* Current or previous use of oral or injectable corticosteroids,
* Have excessive alcohol intake, defined as a daily limit of 30 g (3 drinks) for men and 20 g (2 drinks) for women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To determine liver fat fraction evolution induced by liraglutide and insulin | 12 weeks
  Improvement in liver steatosis defined by change in liver fat fraction as measured by MRI and MR spectroscopy at baseline and 12 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: An Tang, MD, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Tang A, Rabasa-Lhoret R, Castel H, Wartelle-Bladou C, Gilbert G, Massicotte-Tisluck K, Chartrand G, Olivie D, Julien AS, de Guise J, Soulez G, Chiasson JL. Effects of Insulin Glargine and Liraglutide Therapy on Liver Fat as Measured by Magnetic Resonance in Patients With Type 2 Diabetes: A Randomized Trial. Diabetes Care. 2015 Jul;38(7):1339-46. doi: 10.2337/dc14-2548. Epub 2015 Mar 26. PMID 25813773